CLINICAL TRIAL: NCT03498703
Title: Azathioprine in Recurrent Implantation Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Capital Birth Center (Unknown)
Responsible Party: Principal Investigator, Ahmed Reda, Consultant, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FW000372
Record Dates: First submitted 2018-04-07; First posted 2018-04-17 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Recurrent Implantation Failure; In Vitro Fertilization; Intracytoplsmic Sperm Injection
MeSH Terms: interventions — Azathioprine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azathioprine (Experimental)
  Interventions: Drug: Azathioprine Pill
- Control (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Azathioprine Pill — Azathioprine increase pregnancy rate in cases with recurrent implantaion failure
  Arms: Azathioprine
Drug: Placebo Oral Tablet — Placebo tablets
  Arms: Control

SUMMARY:
Azathioprine increase pregnancy rate in patients with recurrent implantation failure

ELIGIBILITY:
Inclusion Criteria:

* age: 20-39
* previous 3 or more failed ivf

Exclusion Criteria:

* intrauterine anomalies
* chronic systemic illness
* chronic pelvic conditions
* sensitivety to azathioprine

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 2 weeks

SECONDARY OUTCOMES:
Side effects | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed H Salama, Study Director — Capital Birth Center
Locations (2):
- Egypt (2):
  - Ain Shams University, Maternity Hospital, Cairo
  - Capital Birth Center, Cairo

IPD SHARING:
Plan to Share IPD: Undecided